CLINICAL TRIAL: NCT06117306
Title: MDMA-assisted Massed Prolonged Exposure for PTSD
Acronym: MDMA-PE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Healing Breakthrough (Unknown)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency); National Center for PTSD (U.S. Federal Agency); White River Junction VA Medical Center (Unknown); Lykos Therapeutics (Industry)
Responsible Party: Principal Investigator, Dr. Leslie Morland, Dr. Leslie Morland, San Diego Veterans Healthcare System
Organization: San Diego Veterans Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVAPT4
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder; MDMA; 3,4-methylenedioxymethamphetamine; Veterans; Prolonged Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized in a stratified 1:1 manner to receive a dose of MDMA (exact doses not disclosed).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Access to the randomization code will be strictly controlled and only available to the un-blinded VA San Diego Research Pharmacist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose A (exact dose not disclosed) (Experimental): Non-medicine sessions of PE + One Medicine Session with 3,4-methylenedioxymethamphetamine (MDMA)
  PE Non-medicine sessions: 12 sessions
  MDMA Medicine session:
  Dose: exact dose not disclosed
  Interventions: Drug: 3,4 Methylenedioxymethamphetamine; Behavioral: Prolonged Exposure
- Dose B (exact dose not disclosed) (Experimental): Non-medicine sessions of PE + One Medicine Session with 3,4-methylenedioxymethamphetamine (MDMA)
  PE Non-medicine sessions: 12 sessions
  MDMA Medicine session:
  Dose: exact dose not disclosed
  Interventions: Drug: 3,4 Methylenedioxymethamphetamine; Behavioral: Prolonged Exposure

INTERVENTIONS:
Drug: 3,4 Methylenedioxymethamphetamine — 1 MDMA session
  Other Names: MDMA
Behavioral: Prolonged Exposure — 12 90-minute PE sessions; initial two sessions both occurring during the first treatment visit, third and fourth sessions occurring during the MDMA session, and the remaining sessions occurring daily or every other day
  Other Names: PE

SUMMARY:
The overall objective of this study is to pilot the VASDHS-adapted Emory MDMA-PE Protocol (aE-MDMA-PE) and assess the effect on clinician-rated PTSD symptoms in veterans who receive different doses of MDMA.

DETAILED DESCRIPTION:
The study is a randomized pilot study that will evaluate the preliminary efficacy, safety, tolerability, and acceptability of the intervention in a sample of U.S. veterans seeking PTSD treatment at the VASDHS. Ten to twenty veterans will be randomized to receive a dose of MDMA (exact range not disclosed) based on the 2-week Emory MDMA-PE Protocol developed by Maples-Keller and Rothbaum. The current protocol will entail massed-PE and the MDMA administration spanning approximately 3-weeks. PE will involve twelve 90-minute sessions with the initial two sessions both occurring during the first treatment visit, the third and fourth sessions occurring during the MDMA session, and the remaining sessions occurring daily or every other day (M-F for two to three weeks).

Following the baseline assessment during Visit 1, participants will begin PE during Visit 2, which will include psychoeducation, rationale for exposure-based treatment, discussion of the SUDS scale, and creating the in vivo exposure hierarchy. Visit 3 will be the Preparatory Session, in which we will provide psychoeducation regarding MDMA's subjective effects and strategies for MDMA-related support. Visit 4 will include the MDMA administration, which will include the third and fourth PE sessions, including the first and second imaginal exposures. Participants will report SUDS at the start and end of imaginal exposure. At the beginning of Visit 5, following a modified version of the MAPS Integration session criteria, the therapist and patient will focus on developing a deeper understanding of insights from the MDMA session and any thoughts or feelings regarding the patient's experience of PTSD and its impact on their life. After the Integration session there will be a break before the PE session. Visits 5-12 will include imaginal exposures and processing of the in-session experience. Imaginal exposures will be recorded, and participants will listen to this recording as homework. Each visit an in vivo exposure will be assigned for homework; all sessions will begin with a check-in that includes reviewing this exposure experience. The post-treatment questionnaire assessment will occur on Visit 13. Participants will complete post-treatment follow-up CAPS-5 clinical interviews remotely approximately 1 week, 2 months, and 4 months after treatment. Following the 2-month follow-up assessment and unblinding, veterans may be offered an optional additional MDMA session and up to three optional additional integration sessions depending on the dose they received.

Participants will be invited to enroll in an optional fMRI (brain imaging) sub-study where, if eligible and interested, they will undergo fMRI brain scans pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be a veteran (age 18-64 years old) who meets criteria for PTSD on the CAPS-5 (severity ≥ 25).
2. Be fluent in speaking and reading English.
3. Are willing to commit to medication dosing, therapy sessions, follow-up sessions, completing evaluation instruments, and all necessary telephone contact
4. Be able to swallow pills.
5. Agree to have study visits audio and/or video recorded, including MDMA session, assessments, and PE sessions, and aware that Independent Rater assessments for PE sessions will occur.
6. Have a contact able to drive the participant home after the MDMA session.
7. Provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
8. Agree to inform the investigators within 48 hours of any new medical conditions or procedures.
9. If able to become pregnant (i.e., assigned female at birth, fertile, following menarche and until becoming post-menopausal unless permanently sterile), must have a highly sensitive negative pregnancy test at study entry and prior to the MDMA session, and must agree to use adequate birth control for 1 month before through 10 days after the MDMA session. Adequate birth control methods include intrauterine device (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e., condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom).
10. Agree to the following lifestyle modifications (described in more detail in Section 3.3 Lifestyle Modifications): comply with requirements for fasting and refraining from certain medications prior to and following the MDMA session, including a possible medication taper if on SSRIs, medications for ADHD, and/or other medications described in the concomitant medications section.
11. Agree not to participate in other PTSD psychotherapy during study treatment.
12. Not enroll in any other interventional clinical trials during the duration of the study, and commit to medication dosing, therapy, and study procedures.
13. At Pre-Screening, have at least moderate PTSD symptoms in the last month based on PCL-5 total score of 40 or greater (index).
14. May have well-controlled hypertension that has been successfully treated with anti- hypertensive medicines if they pass additional screening to rule out underlying cardiovascular disease.
15. May have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
16. May have alcohol or substance use disorder if participant is not in withdrawal or requiring detox. Participants must have a plan, agreed upon by investigator, therapy team, and study physician, to reduce use of alcohol or other substances and to manage symptoms without self-medicating. Enrollment will require that, in the judgment of the investigator, therapy team, and study physician, the plan for decreasing substance use is realistic and has a good chance of succeeding in order to prevent substance use from impacting the safety or effectiveness of the investigational treatment. Veterans will also be subject to a urine toxicology drug screening prior to enrollment and before the MDMA session.
17. May have a history of or current Diabetes Mellitus (Type 2) if additional screening measures rule out underlying cardiovascular disease, if the condition is judged to be stable on effective management, and with approval by the study physician.
18. May have hypothyroidism if taking adequate and stable thyroid replacement medication.
19. May have a history of, or current, glaucoma if approval for study participation is received from an ophthalmologist.

Exclusion Criteria:

1. Are not able to give adequate, written informed consent.
2. Are currently engaged in compensation and pension (C&P) litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders.
3. Are likely, in the investigator's opinion and via assessment period, to be re- exposed to their index trauma or other significant trauma, lack social support, or lack a stable living situation.
4. Have used Ecstasy (material represented as containing MDMA) or have participated in an MDMA clinical trial.
5. Have a positive screen for amphetamine or cocaine.
6. Have any current problem which, in the clinical opinion of the investigator and study physician, might interfere with participation due to it impacting the patient's safety and/or ability to participate in the protocol.
7. Have hypersensitivity to any ingredient of the IMP (Investigational Medicinal Product).
8. Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment.
9. Have dementia.
10. Have a history of or a current primary psychotic disorder assessed via the DIAMOND and clinical interview.
11. Have a history of or current Bipolar 1 disorder, Bipolar 2 disorder, or manic episode assessed via the DIAMOND and clinical interview.
12. Have a current eating disorder with active purging assessed via DIAMOND and clinical interview.
13. Have current major depressive disorder with psychotic features assessed via DIAMOND.
14. Have a current panic disorder assessed via the DIAMOND
15. Have a history of amphetamine or cocaine substance use disorder
16. Have a current alcohol or substance use disorder other than caffeine or nicotine that the investigators, therapy team, and/or study physician judge to be a safety concern for enrollment in the study or that could interfere with the therapeutic process or with other aspects of study participation. Any participant who is not able to agree or adhere to a plan to reduce use and manage symptoms will not be enrolled. Individuals endorsing severe symptoms of an active alcohol use disorder (AUDIT >8 for men, >6 for women) or of an active substance use disorder (DUDIT >6 for men, >2 for women) will be evaluated by the study PI and/or physicians to determine if they should be excluded.
17. Present with current serious suicide risk, as determined through psychiatric interview, responses to C-SSRS (scores of four or greater), and clinical judgment of the investigator; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior, in the judgment of the investigator, will not be enrolled. Any participant presenting with the following on the pre-screen C-SSRS will be excluded:

    1. Suicidal ideation score of 4 or greater within the last 6 months of the assessment at a frequency of once a week or more.
    2. Any suicidal behavior, including suicide attempts or preparatory acts, within the last 6 months of the assessment. Participants with non-suicidal self- injurious behavior may be included if approved by the study physician.
18. Would present a serious risk to others as established through clinical interview and if necessary, discussion with treating psychiatrist.
19. Require ongoing concomitant therapy with a psychiatric medication other than the exceptions described in protocol section on Concomitant Medications.
20. Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate. This includes, but is not limited to, a history of myocardial infarction, cerebrovascular accident, or aneurysm. Participants with other mild, stable chronic medical problems may be enrolled if the study physician and PI agree the condition would not significantly increase the risk of MDMA administration or be likely to produce significant symptoms during the study that could interfere with study participation or be confused with side effects of the IMP. Examples of stable medical conditions that could be allowed include, but are not limited to Human Immunodeficiency Virus (HIV) infection, Gastroesophageal Reflux Disease (GERD), etc. Any medical disorder judged by the investigator to significantly increase the risk of MDMA administration by any mechanism would require exclusion.
21. Have a diagnosis of uncontrolled hypertension defined by the American Heart Association as repeated readings of ≥ 140 millimeters of Mercury [mmHg] systolic or ≥ 90 mmHg diastolic.
22. Have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease.
23. Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
24. Have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening. Participants with a history of atrial fibrillation, atrial tachycardia, atrial flutter or paroxysmal supraventricular tachycardia or any other arrhythmia associated with a bypass tract may be enrolled only if they have been successfully treated with ablation and have not had recurrent arrhythmia for at least one year off all antiarrhythmic drugs and confirmed by a cardiologist.
25. Have a marked Baseline prolongation of QT/QTc interval. For purposes of eligibility, this is defined as repeated demonstration of a QT interval corrected using Fridericia's formula [QTcF] >450 milliseconds [ms].
26. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
27. Require use of concomitant medications that prolong the QT/QTc interval during Sessions. Refer to protocol section on Concomitant Therapy.
28. Have symptomatic liver disease or have repeated significant liver enzyme elevations on labs.
29. Have history of hyponatremia or hyperthermia.
30. Have a BMI of 18.5 or less.
31. Are pregnant or nursing or are able to become pregnant and are not willing/able to practice an effective means of birth control.
32. Have engaged in ketamine-assisted therapy or used ketamine within 12 weeks of enrollment.
33. Have any preexisting condition affecting renal functioning.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinician-rated PTSD symptoms | Baseline - 4-months post-treatment
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a 20-item diagnostic interview administered by trained evaluators to assess PTSD in a participant. Based on DSM-5 diagnostic criteria, evaluators ask about the severity of four PTSD-related symptom clusters: re-experiencing, avoidance, negative alterations in cognition and mood, and alterations in arousal and reactivity. The evaluator rates responses on a 5-point Likert scale (0 = Absent to 4 = Extreme/Incapacitating). Total scores range from 0 to 80 with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Self-reported PTSD symptoms | Baseline - 4-months post-treatment
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms. Participants indicate how much distress they have experienced due to symptoms on a five-point Likert-type scale (1=Not at all to 5=Extremely). Total scores range from 0 to 80, with higher scores indicating more severe PTSD symptoms.
Depressive Symptoms | Baseline - 4-months post-treatment
  The Patient Health Questionnaire 9 (PHQ-9) is a 9-item self-report measure of depressive symptoms. The PHQ-9 screens for major depression, with a score of 10 or above indicative of a possible major depressive episode, and it provides a measure of severity of these symptoms.
Functioning | Baseline - 4-months post-treatment
  The Brief Inventory of Psychosocial Functioning (B-IPF) is a brief version of the Inventory of Psychosocial Functioning (IPF) that measures functioning impairment across seven domains: intimate relationships, family and parenting, friendships, work, socializing, education, and self-care over the past 30 days. Total scores, ranging from 0 to 100, are calculated as the sum score divided by the total possible score multiplied by 100, with higher scores indicating greater impairment in functioning.
Sleep | Baseline - 4-months post-treatment
  The Pittsburgh Sleep Quality Index (PSQI) measures sleep quality over the past 1-month using 19 items in a self-report questionnaire format. The scale has seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Items are rated on a combination of Likert scales from 0 to 3 and open- ended questions that are later converted to scaled scores. Higher total scores indicate greater sleep disturbance.
Safety/Suicidality | Baseline - 4-months post-treatment
  The C-SSRS is a clinician-administered measure of suicidal behavior devised to detect potential suicidal thoughts or behaviors during a clinical trial. It consists of a Baseline version and a Since Last Visit version that assess suicidal ideation, ideation intensity, and behavior.
Sexual Functioning | Baseline - 4-months post-treatment
  The CSFQ-14 is a 14-item self-report scale that evaluates sexual functioning. The measure has five subscales: pleasure, desire/frequency, desire/interest, arousal/excitement, and orgasm/completion. All items are scored on 5-point scales with varying response options. Higher total scores indicate better sexual functioning. The CSFQ-14 has corresponding assigned-male-at-birth and assigned-female-at-birth versions.
Moral Injury | Baseline - 4-months post-treatment
  The MIDS is a two-part self-report measure that examines potentially morally injurious events (PMIEs) exposure and moral injury symptoms in the past month. The first part of the scale uses 6 items to measure exposure to and bothersomeness of PMIEs through a 5-point Likert scale (0=Not at all to 4=Extremely). The second part of the scale includes a series of open-ended questions to select and describe the most distressing PMIE. Respondents then complete 18 items that are scored on 5-point Likert scales to indicate their cognitive, emotional, behavioral, social, and religious or spiritual reactions to the PMIE that they find the most distressing. Higher summed score indicates more severe moral distress.
Adverse Childhood Experiences | Baseline
  Measured using the Adverse Childhood Events Scale (ACES). The ACES is a 10-item self-report survey that asks about childhood stress. Participants indicate exposure to different kinds of abuse with yes/no responses, and answer "1" if the abuse happened often. Higher scores indicate greater exposure to childhood stressors.
Posttraumatic Growth | Baseline - 4-months post-treatment
  Measured using the Posttraumatic Growth Inventory (PTGI). The PTGI is a 21-item self-report measure that asks about level of posttraumatic growth across 5 subscales in adults who have experienced trauma. Participants respond using a 6-point Likert scale (1=I did not experience this change as a result of my crisis, to 6=I experienced this change to a very great degree as a result of my crisis).Total scores range from 1-126.
Anger | Baseline - 4-months post-treatment
  The STAXI-2 is a 57-item self-report measure that assesses the respondent's experience, expression, and control of anger. The measure includes six scales; for the purpose of this study, only the state anger state anger (i.e., the intensity of anger at the time of completing the scale; 15 items) and trait anger (i.e., whether the person has an overall angry temperament; 10 items) scales will be used, for a total of 25 items. All items are rated on a scale from 1 (Almost never) to 4 (Almost always). Both scales are scored by summing responses to each item, with higher scores indicating higher state and/or trait anger. Ranges are 15-60 for the state scale and 10-40 for the trait scale.
Well Being | Baseline - 4-months post-treatment
  Measured using the Well-Being Signs (WBS). The WBS is a 3-item self-report measure examining psychosocial well-being. All items are rated on a scale from 0 to 10. An average score is calculated based on the ratings for each question. Higher scores indicate better psychosocial well-being.

OTHER OUTCOMES:
Satisfaction with Care | 1 week post-treatment
  The Client Satisfaction Questionnaire - 8-item version (CSQ-8) is an 8-item survey of patient satisfaction with healthcare or services that they are receiving. Items are rated on Likert scales from 0 to 3 with varying response options based on the question. Questions address varying aspects of satisfaction with care. Higher scores indicate higher satisfaction.
Acceptability of Care | 1 week post-treatment
  Audiotaped Qualitative Interview
Treatment Expectations | Baseline, Visit 3
  Measured using the Stanford Expectations of Treatment Scale (SETS). The SETS is a 10-item self-report questionnaire that assesses a patient's feelings about their upcoming treatment. The first 6 items are rated on a 7-point Likert scale (1=strongly disagree, to 7=strongly agree). Items 7-9 are open-ended. Item 10 is a yes/no response. The scale yields a score for positive expectancy and negative expectancy.
Trauma Exposure | Baseline
  Measured using the Life Events Checklist for DSM-5 (LEC-5). The LEC-5 is a 17-item self-report survey that asks about exposure to potentially traumatic events. Participants indicate the type of exposure for each event (Happened to me, Witnessed it, Learned about it, Part of my job, Not sure, Doesn't apply).

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Morland, Psy.D., Principal Investigator — San Diego Veterans Affairs Health System
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided